CLINICAL TRIAL: NCT04768478
Title: The Use of Cannabidiol (CBD) in Pain Reduction and Opioid Use After Ankle and Tibia Fracture Open Reduction and Internal Fixation. A Double-Blind, Randomized Control Study
Brief Title: CBD for Pain Reduction and Opioid Use After Ankle and Tibia Fracture ORIF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: there was no funding to begin the study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-00069
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Ankle Fractures; Tibia Fracture
Keywords: Cannabidiol
MeSH Terms: conditions — Ankle Fractures; Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Active Comparator)
  Interventions: Drug: CBD
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — 25mg CBD ODTs (orally disintegrating tablet), with instructions to take CBD tablets t.i.d. (total of 50mg per dose t.i.d.) to be administered with routine post-operative pain management
  Arms: Cannabidiol (CBD)
Drug: Placebo — Visually indistinguishable placebo ODTs, with instructions to take two tablets t.i.d., to be administered with routine post-operative pain management
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of administering CBD to control post-operative pain in patients undergoing ankle fracture open reduction and internal fixation, tibial plafond (pilon) open reduction and internal fixation, tibial shaft repair (open reduction internal fixation or intramedullary nail fixation), or tibial plateau open reduction and internal fixation. Secondly, the purpose is to evaluate the effectiveness of CBD in comparison with opioid therapy for post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an ankle fracture open reduction and internal fixation (medial malleolus, lateral malleolus, posterior malleolus, and/or syndesmosis repair), tibial plafond (pilon) open reduction and internal fixation, tibial shaft repair (open reduction internal fixation and intramedullary nail fixation), or tibial plateau open reduction and internal fixation
* Patients ages 18-75, inclusive
* Female patients must be currently practicing effective forms of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (less than 1% per year) when used consistently and correctly
* Male patients must be using an effective form of contraception

Exclusion Criteria:

* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Older than 75 years of age
* Any patient considered a vulnerable subject: pregnant women or fetuses, children, cognitively impaired adults, prisoners
* History of cannabis abuse or dependence
* History of coagulation abnormalities and thromboembolic disease or current abnormal coagulation test values
* History of stroke or acute coronary syndromes within 3 months before surgery
* Abnormal coagulation profile
* Renal failure (serum creatinine > 250 μmol/L [2.83 mg/dL]) or liver cirrhosis
* Patients that have been on pre-operative opioid management for any reason
* Patients meeting the DSM-V for major psychiatric illness, such as bipolar disorder
* Patients diagnosed with major depression, psychosis, or substance abuse disorder
* Patients with current or a history of suicidal ideation
* Breastfeeding females
* Patients with clinically significant illness, including cardiovascular disorders
* Clinically significant lab abnormalities
* Abnormal LFTs
* Patients with major neurological disorders, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain/head injury, or seizures
* Patients with moderate (Child-Pugh B) and severe hepatic impairment (Child-Pugh C).
* Patients taking moderate or strong inhibitors of CYP3A4 and CYP2C19 concomitantly
* Patients taking strong CYP3A4 and CYP2C19 inducers concomitantly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Score on Pain Visual Analog Scale (VAS) | Day 2 Post-Surgery
  Pain severity scores at rest will be assessed by use of a visual analog scale (VAS; total range = 0-10; 0 = no pain, 10 = worst pain imaginable)
Score on Pain Visual Analog Scale (VAS) | Day 7 Post-Surgery
  Pain severity scores at rest will be assessed by use of a visual analog scale (VAS; total range = 0-10; 0 = no pain, 10 = worst pain imaginable)
Score on Pain Visual Analog Scale (VAS) | Day 14 Post-Surgery
  Pain severity scores at rest will be assessed by use of a visual analog scale (VAS; total range = 0-10; 0 = no pain, 10 = worst pain imaginable)
Level of Nausea Using VAS | Day 2 Post-Surgery
  Any nausea experienced by the patients will be recorded by use of a VAS (total range = 0-10; 0 = no nausea, 10 = worst nausea imaginable)
Level of Nausea Using VAS | Day 7 Post-Surgery
  Any nausea experienced by the patients will be recorded by use of a VAS (total range = 0-10; 0 = no nausea, 10 = worst nausea imaginable)
Level of Nausea Using VAS | Day 14 Post-Surgery
  Any nausea experienced by the patients will be recorded by use of a VAS (total range = 0-10; 0 = no nausea, 10 = worst nausea imaginable)

SECONDARY OUTCOMES:
CBD Consumption | Day 2 Post-Surgery
  Patient self report
CBD Consumption | Day 7 Post-Surgery
  Patient self report
CBD Consumption | Day 14 Post-Surgery
  Patient self report
Opioid Consumption | Day 2 Post-Surgery
  Patient self report
Opioid Consumption | Day 7 Post-Surgery
  Patient self report
Opioid Consumption | Day 14 Post-Surgery
  Patient self report
Patient Satisfaction Score | Day 14 Post-Surgery
  Patients will record their satisfaction with their management, on a 0-10 scale. The higher the score, the higher the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Leucht, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Orthopedic Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Philipp.Leucht@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.